CLINICAL TRIAL: NCT01278706
Title: Comparing Timing and Number of Endometrial Biopsies in IVF Treatment and Identifying Biochemical Markers to Predict Endometrial Receptivity
Brief Title: Endometrial Biopsy Protocol for In Vitro Fertilization (IVF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Amihai Barash M.D. IVF Unit Director, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kmc110154CTIL
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-12

CONDITIONS: Infertility; Recurrent Implantation Failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- no treatment (No Intervention)
- one biopsy, proliferative phase (Experimental)
  Interventions: Procedure: endometrial biopsy/ies
- one biopsy, secretory phase (Experimental)
  Interventions: Procedure: endometrial biopsy/ies
- two biopsies (Experimental)
  Interventions: Procedure: endometrial biopsy/ies

INTERVENTIONS:
Procedure: endometrial biopsy/ies — performing office endometrial biopsy with a disposable sterile catheter
  Arms: one biopsy, proliferative phase; one biopsy, secretory phase; two biopsies

SUMMARY:
Endometrial biopsy has been shown to improve IVF pregnancy and live birth rates. The optimal time of performing the biopsy is yet to be established.

In this study, the investigators will compare different temporal timing of the biopsies with regards to the menstrual cycle and their affect on the success rates of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* normal menstrual cycle
* between 1-6 previous failed IVF cycles
* normal hormonal profile

Exclusion Criteria:

* intrauterine procedure in last 3 months
* hydrosalpinx
* intrauterine lesion /malformation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy rates | 2 years

SECONDARY OUTCOMES:
live birth rates | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Kaplan Medical Center, IVF Unit, Rehovot
  - Weizmann Institute of Science, Rehovot